CLINICAL TRIAL: NCT05467488
Title: Ultraviolet A and Ultraviolet C Light-induced Effects on Dental Implant Stability
Brief Title: Light-induced Effects on Dental Implant Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Abdul Mueed Zaigham (Other)
Responsible Party: Sponsor-Investigator, Prof. Abdul Mueed Zaigham, Professor, CMH Lahore Medical College and Institute of Dentistry
Organization: CMH Lahore Medical College and Institute of Dentistry (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32/ERC/CMH/LMC
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Missing Teeth
Keywords: dental implants
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non irradiated implants (group A) (No Intervention)
- UVA irradiated group (group B) (Active Comparator)
  Interventions: Procedure: photofunctionalization
- UVC irradiated group (group C) (Active Comparator)
  Interventions: Procedure: photofunctionalization

INTERVENTIONS:
Procedure: photofunctionalization — UVA and UVC photofunctionalization of dental implants
  Arms: UVA irradiated group (group B); UVC irradiated group (group C)

SUMMARY:
Until now, limited research has observed the stability of photo functionalized sandblasted acid-etched (SLA) titanium implants. The study includes a sample size of sixty otherwise healthy patients with implant replacement, comparing nonirradiated, irradiated UVA and UVC titanium implants. It was an interventional study with a sample size divided into three groups using simple randomization. Patients with nonirradiated dental implants make the control group A with UVA and UVC dental implants forming groups B and C, respectively. Before functional loading, implant stability was measured on days zero and eight weeks. SPSS 26.0 is used for data analysis. The data for implant stability quotient (ISQ) levels and osseointegration speed index (OSI) were presented as mean ± SD for each group. The effect of UVA and UVC on ISQ2 compared with the baseline ISQ was done by applying multiple simple regression analysis models, whereas the distinction between UVA and UVC was made through a t-test. p ≤ 0.05 was kept statistically significant. The implants irradiated with UVA significantly affected ISQ levels compared to other groups.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients with age > 20 with at least one tooth or more missing

Exclusion Criteria:

-

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
ISQ measurement through Ostelltm Mentor device | eight months
  The Ostelltm device was initially calibrated using a test peg called the ISQ. A smart peg was used for assessment. The smart peg tightened with 5 Ncm torque is then mounted on implant fixture and the transducer connected perpendicular to the implant . The measuring probe is brought closer to the smart peg without touching it. A beeping sound displays the reading on the monitor. Two successive readings are taken mesiodistally along the jaw and buccolingually perpendicular to the jaw .The RFA measurements taken twice during implant treatment are recorded. All the ISQ values were recorded from one to hundred and a mean was taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Dentistry; CMH Lahore Medical College, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided